CLINICAL TRIAL: NCT02152449
Title: Impact on Functional Status of Early Oral Nutritional Supplementation (ONS) in Amyotrophic Lateral Sclerosis (ALS) Patients
Brief Title: Oral Nutritional Supplementation in Amyotrophic Lateral Sclerosis (ALS) Patients
Acronym: NUTRALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Laboratoires NUTRICIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I12025
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2019-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group: systematic advice on swallowing, plus:
  * If no weight loss compared to usual weight: no intervention
  * if weight loss <5%: advice on a fat- and protein-enriched diet
  * if weight loss ≥5%: advice on a fat- and protein-enriched diet + 1 unit of ONS/day per os
- oral nutritional supplementation (Experimental): Experimental "ONS" Group: systematic advice on swallowing + systematic advice on a fat- and protein-enriched diet, plus:
  * if no weight loss compared to usual weight: 1 ONS/day per os
  * if weight loss <5% compared to usual weight: 2 ONS/day per os
  * if weight loss ≥5% compared to usual weight: 3 ONS/day per os
  Interventions: Dietary Supplement: Oral nutritional supplementation

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplementation
  Other Names: Fortimel Compact Protein ®; Fortimel Crème®
  Arms: oral nutritional supplementation

SUMMARY:
The purpose of this study is to determine whether an early oral nutritional supplementation (ONS) in amyotrophic lateral sclerosis (ALS) patients is effective on the treatment of this rapidly progressive disease.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rare neurodegenerative disease with a median age at time of diagnosis of 65 years. In France, the incidence ranges between 1.5 and 2.5/100 000 person-year of follow-up. The disease is related to progressive degeneration of motor neurons in the two voluntary motor pathways. It is a very debilitating disease, particularly in terms of autonomy and respiratory function. Its prognosis is poor, with constant worsening during the follow-up, leading to death with a median survival of 24 months after diagnosis. ALS patients are at risk of malnutrition in the short and medium term, because of several factors limiting or stopping food intake, such as functional disability, and swallowing or breathing disorders. The disease is also accompanied in 50-60% of cases by an abnormal increase in energy expenditure (hypermetabolism), causing added weight loss. Previous studies have shown that malnutrition is an independent negative prognostic factor for survival. Besides, at time of diagnosis, 36% of patients have already lost more than 5% of their usual weight. Such a weight loss has been shown to be associated with a 2 fold increased risk of dying, after adjustment for other known prognostic factors. Moreover, patients with a higher fat body mass during the course of the disease have a significant increased survival; and higher levels of serum cholesterol and/or triglycerides are favourable factors for survival. The recommendations for the management of ALS patients, published by French and International groups of experts, have suggested the use of oral nutritional supplementation if food intake does not cover the patient's requirements.

We propose that Oral Nutritional Supplementation (ONS) should be used (i) systematically and (ii) earlier (as early as the time of diagnosis) in order to enable patients to maintain proper nutritional status.

Such an intervention could delay the progression of the disease if the metabolic disorders in ALS are not solely the result of progression of the disease, but are implicated in its course and outcome.

This is a parallel randomized study aimed To assess the benefits of early oral nutritional supplementation (ONS) on neurological functional status evaluated by the slope of the revised ALS Functional rating Scale (ALSFRS-R) between inclusion (T0) and T0+6 months in newly diagnosed ALS pati

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age, diagnosed with ALS (<2 months before inclusion) according to Airlie House criteria : definite, probable, or probable laboratory supported;
* Time between first symptoms and diagnosis less than 18 months
* Sporadic or familial cases
* Patient agreement to be followed in a given ALS centre during the duration of the study
* Patients with a loss of at least 1 point in 3 items of the ALSFRS-R rating scale or with a loss of at least 2 points in 2 items of the ALSFRS-R rating scale
* Patients who signed the informed consent form

Exclusion Criteria:

* Associated dementia or inability to understand the requirements of the protocol.
* No helper
* ONS already begun
* Artificial nutrition: enteral or parenteral nutrition
* Known hypersensitivity to components of ONS
* Absence of treatment with Riluzole (RILUTEK®)
* Patient under guardianship or curatorship
* Participation in another research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change in the ALSFRS-R slope between T0 and T0+6 months | Month 6
  Change in the ALSFRS-R slope between T0 and T0+6 months (ALSFRS-R will be assessed by an examiner blinded to the intervention group).

SECONDARY OUTCOMES:
Combined assessment of Function and Survival (CAFS) | Mont 3 and month 6
  Combined assessment of Function and Survival (CAFS)
Body Mass Index and of Fat Mass. | Day 1, month 3, months 6:
  Nutritional status will be evaluated by means of Body Mass Index and of Fat Mass.
  Measurement will be performed at T0, T0+3 months and T0+6 months:

CONTACTS AND LOCATIONS:
Overall Officials: Philippe COURATIER, MD, Principal Investigator — CHU Limoges
Locations (1):
- Service de Neurologie, Limoges, France